CLINICAL TRIAL: NCT02876718
Title: Xarelto Evidence in Real Life of Patients Preference and Satisfaction Study.
Brief Title: Xarelto Evidence in Real Life of Patients' Preference and Satisfaction Study
Acronym: X-PRESS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18728
Record Dates: First submitted 2016-07-22; First posted 2016-08-24 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban, BAY59-7939: It is a single-arm study in which only patients who switched from a VKA to a NOAC treatment will be included.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY 59-7939) — No specified dosing or dosage in the study. The treatment decision falls within current practice and the prescription of the medicines is clearly separated from the decision to include the patient in the study.

SUMMARY:
The main objective of the study is to assess preferences of Non Valvular Atrial Fibrillation (NVAF) patients towards different options of an anticoagulation treatment.

Patient preferences for anticoagulant treatment attributes (convenience attributes only), based on a Discrete Choice Experiment(DCE) interview will be elicited and the impact of switching from Vitamin K Antagonist(VKA) to Xarelto® on Atrial Fibrilation(AF) patient treatment satisfaction will be documented, measured by score differences of the Anti-Clot Treatment Scale (ACTS) score in patients switching from VKA to Rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 20 years of age (legal age limit in Taiwan) with a confirmed diagnosis of AF (non-valvular).
* Treatment with VKA for at least 6 weeks.
* Decision to initiate treatment with Rivaroxaban has been made as per investigator's routine treatment practice.
* Written informed consent of the patient.
* Wilingness and capability to conduct two F2F interviews.

Exclusion Criteria:

* Contraindications to the use of Rivaroxaban as outlined in the local product information .
* Concomitant treatment with any other anticoagulants.
* Participation in another study (clinical intervention/observational) within the 3 months prior to enrollment.
* Patients participating in an investigational program with interventions outside of routine clinical practice.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients will be included in this study. Participating centers are either primary care practices, internal medicine specialist practices or out-patient sites/out-patient clinics
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Patient preferences for anticoagulant treatment attributes (utility values obtained in Logit/Probit estimates) | At 3 months
  The preferred attributes will be assessed by a questionnaire following a discrete choice experimental design.

SECONDARY OUTCOMES:
Change of the Anti-clot treatment scale (ACTS) benefit and burden score from baseline (on VKA) to 3 months (on Xarelto) | At 0 month and at 3 months
  ACTS = Anti Clot treatment Scale is a questionnaire of 17 items (13 items on burden of treatment and 4 items on the benefits of treatment)
AF symptoms as measured by European Heart Rhythm Association (EHRA) symtoms (both severity and frequency) | At 3 months
Reasons for switch from VKA to Xarelto | At 0 month
  The reasons are selected by the participant out of a qualitative list of reasons for switch from VKA to Xarelto.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Taiwan